CLINICAL TRIAL: NCT04542356
Title: Efficacy and Safety of PEGylated Recombinant Human Granulocyte Stimulating Factor in the Prevention of Neutropenia During Concurrent Chemoradiotherapy for Cervical Cancer
Brief Title: Study on the Efficacy and Safety of PEG-rhG-CSF in Preventing Neutropenia During Concurrent Chemoradiotherapy of Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Associated Director, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CQGOG0104
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; concurrent chemoradiotherapy; neutropenia; PEG-rhG-CSF
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): patients used 6 mg PEG-rhG-CSF prophylactically after chemotherapy
  Interventions: Drug: PEG-rhG-CSF
- control group (Placebo Comparator): patients did not use PEG-rhG-CSF for prevention and were given 5 ug/kg rhG-CSF when ANC<1✕109/L
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — During the concurrent chemoradiotherapy, a single subcutaneous injection of 6 mg PEG-rhG-CSF was given to the patient 2 hours after radiotherapy on the first day after the end of chemotherapy. Blood tests were performed weekly, if the patient's neutrophils were less than 1.0 × 109 / L during radiotherapy, rhG-CSF was given as a remedial treatment. If fever occurs, antibiotics were given promptly.
  Arms: experimental group
Drug: rhG-CSF — Blood tests were performed weekly, if the patient's neutrophils were less than 1.0 × 109 / L during radiotherapy, rhG-CSF was given as a remedial treatment. If fever occurs, antibiotics were given promptly.
  Arms: control group

SUMMARY:
This randomized controlled prospective study aims to explore the efficacy and safety of using (PEGylated Recombinant Human Granulocyte Stimulating Factor) PEG-rhG-CSF to prevent neutropenia during concurrent chemoradiotherapy of paclitaxel and cisplatin (TP) regimen for cervical cancer. To find out the best time to use PEG-rhG CSF, and to explore investigate the effect of PEG-rhG-CSF on long-term bone marrow function in the process of concurrent chemoradiotherapy, and finally to explore the clinical feasibility of using PEG-rhG-CSF to prevent neutropenia during concurrent chemoradiotherapy of TP regimen for cervical cancer.

DETAILED DESCRIPTION:
Study design: In this prospective, single-center, randomized controlled study, patients with locally advanced cervical cancer are randomly divided into two groups. Patients in the experimental group will receive PEG-rhG-CSF 6mg prevention during concurrent chemoradiotherapy, whereas the control group do not use PEG-rhG-CSF for prevention. When the patient's ANC is less than 1✕109/L, 5μg/kg rhG-CSF will be given for treatment until the ANC returned to 2✕109/L.

Case selection: patients with IIb-IIIb cervical cancer, squamous cell carcinoma confirmed by histopathology, and three-week regimen of paclitaxel and carboplatin with Concurrent Radiotherapy.

Primary end point: incidence and duration of grade 3/4 neutropenia in patients. Secondary endpoints: 1) Incidence of febrile neutropenia (FN); 2) the rate of postponement of the course of radiotherapy, reduction in chemotherapy dose and postponement of the course of chemotherapy; 3) Changes of bone marrow function in patients 3 months and 6 months after radiotherapy.

Safety assessment: laboratory safety testing, including platelet count and hemoglobin. Evaluation of adverse events: infection, neutropenic fever, bone pain, etc.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old;
* Patients with cervical cancer who have not undergone surgery for initial treatment, the international union of gynecology and obstetrics (FIGO) stage IIb-IIIb; Squamous cell carcinoma diagnosed by histopathology.
* The expected survival time was more than 8 months; the Eastern Cooperative Oncology Group (ECOG) performance status score≤1;
* Bone marrow hematopoietic function is normal before treatment (ANC≥1.8×109/L, PLT≥100×109/L, Hb≥90g/L, WBC≥4.0×109/L);
* No obvious abnormality in the ECG examination, and no obvious cardiac dysfunction;
* All patients must agree to take effective contraceptive measures during the study period and within 6 months after stopping treatment, and women of childbearing age must have a negative urine pregnancy test prior to treatment administration;
* The subjects voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

* Those who refuse to accept PEG-rh-G-CSF;
* Currently conducting clinical trials of other drugs;
* Uncontrolled infection before treatment, body temperature ≥ 38℃;
* Chronic diseases of the heart, kidney, liver or other important organs;
* Patients with severe uncontrolled diabetes;
* Pregnant or lactating female patients;
* Persons with allergic diseases or allergic constitution, or allergic to this product or other biological products derived from genetically engineered E. coli;
* Suspected or confirmed drug, substance or alcohol abuse;
* Severe mental or neurological disorders that affect informed consent and/or adverse reaction presentation or observation;
* HIV-positive people;
* Patients requiring radiation therapy for the retroperitoneal or inguinal region.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 3-4 neutropenia | 2 months
  Incidence of Grade 3-4 neutropenia
Duration of grade 3-4 neutropenia | 2 months
  Duration of grade 3-4 neutropenia

SECONDARY OUTCOMES:
Incidence of febrile neutropenia (FN) | 2 months
  Incidence of febrile neutropenia (FN)
the rate of postponement of the course of radiotherapy | 2 months
  the rate of postponement of the course of radiotherapy
reduction in chemotherapy dose | 2 months
  reduction in chemotherapy dose
postponement of the course of chemotherapy | 2 months
  postponement of the course of chemotherapy
Changes of bone marrow function in patients 3 months and 6 months after radiotherapy | 6 months
  Changes of bone marrow function in patients 3 months and 6 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cartmell MP, Ziegler SW, Neill DS. On the performance prediction and scale modelling of a motorised momentum exchange propulsion tether[J]. Gynecol Oncol, 2003, 654 (1): 571-579.
- [Background] Liu Y, Zhang X, An S, Wu Y, Hu G, Wu Y. Pharmacokinetics of neamine in rats and anti-cervical cancer activity in vitro and in vivo. Cancer Chemother Pharmacol. 2015 Mar;75(3):465-74. doi: 10.1007/s00280-014-2658-7. Epub 2015 Jan 1. PMID 25552400
- [Background] Saha A, Chaudhury AN, Bhowmik P, Chatterjee R. Awareness of cervical cancer among female students of premier colleges in Kolkata, India. Asian Pac J Cancer Prev. 2010;11(4):1085-90. PMID 21133629
- [Background] Moore TD，Patel T，et al．A sir pesfligrastim dose per cycle supports dose-dense(q14d)CHOP-R in patients with non Hodgkin's lymphoma[J]．Proc Am Soc Hematol，2003，102(11): 2365．
- [Background] Lokich J. Same-day pegfilgrastim and chemotherapy. Cancer Invest. 2005;23(7):573-6. doi: 10.1080/07357900500276899. PMID 16305982
- [Derived] Zou D, Guo M, Zhou Q. A clinical study of pegylated recombinant human granulocyte colony stimulating factor (PEG-rhG-CSF) in preventing neutropenia during concurrent chemoradiotherapy of cervical cancer. BMC Cancer. 2021 Jun 2;21(1):661. doi: 10.1186/s12885-021-08364-9. PMID 34078317